CLINICAL TRIAL: NCT05222581
Title: Engineering Evaluation of a Breast Pump Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Momtech Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: MOMI-001
Record Dates: First submitted 2022-01-11; First posted 2022-02-03 (Actual); Last update posted 2025-05-09 (Actual); Status verified 2025-05

CONDITIONS: Healthy; Breast Pumping
MeSH Terms: conditions — Breast Milk Expression

STUDY DESIGN:
Intervention Model Description: Prototype breast shield designs for the Freedom Double Electric Breast Pump with <10 subjects per breast shield design. The study sample size is appropriate for a small feasibility study evaluating design concepts because there are several breast shield designs being evaluated with a small number of subjects per design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Prototypes of Breast Shield and Freedom Double Electric Breast Pump (Experimental): Prototypes of breast shield and Freedom Double Electric Breast Pump
  Interventions: Device: Prototypes of breast shield and Freedom Double Electric Breast Pump

INTERVENTIONS:
Device: Prototypes of breast shield and Freedom Double Electric Breast Pump — Prototypes of breast shield and Freedom Double Electric Breast Pump.

SUMMARY:
This research involves feasibility testing of design concepts to support device development of an electric breast pump. The purpose is to evaluate a prototype device for feasibility purposes and not health outcomes.

DETAILED DESCRIPTION:
This engineering evaluation involves the voluntary participation of healthy adult lactating women for feasibility testing of breast shield designs. Participants will be asked to rate the breast shield design for fit, comfort, and the ease of use. In addition, participants will be asked to rate a comparison of the device relative to their experiences with their current commercial breast pump and breastfeeding their baby.

ELIGIBILITY:
Inclusion Criteria:

* History of good health
* Currently lactating and planning to continue breastfeeding for the next 3 to 4 months
* Currently using a commercial electric breast pump at least several times a week
* Sufficient milk supply for one missed infant feeding per device testing visit
* Willing to attend five device testing visits over 3 to 4 months
* Willing to be video recorded during device testing
* Willing to discard milk collected during testing

Exclusion Criteria:

* No active breast or nipple injury, breast inflammation or infection, or nipple piercing
* No prior history of breast implant, reduction or reconstruction surgery
* Not currently pregnant

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2024-06-01 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Breast shield comfort | 1 day (Single timepoint)
  Rate comfort of device by Questionnaire
Breast shield fit | 1 day (Single timepoint)
  Rate fit of device by Questionnaire
Breast shield ease of use | 1 day (Single timepoint)
  Rate ease of use of device by Questionnaire

SECONDARY OUTCOMES:
Volume of milk expressed | 1 day (Single Timepoint)
  Rate volume of milk expressed with device by Questionnaire
Participant comparison of device to current commercial breast pump | 1 day (single timepoint)
  Rate comparison of device to current breast pump experience by Questionnaire
Participant comparison of device to breastfeeding | 1 day (single visit)
  Rate comparison of device to breastfeeding experience by Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ashley Wofford Leong, MD, Principal Investigator — Independent Physician
Locations (1):
- Blur Product Development, Cary, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No